CLINICAL TRIAL: NCT01621997
Title: Retraining Via Operation Inspection or Verbal Education vs Usual Care on the Prevention of Peritonitis in Peritoneal Dialysis
Brief Title: Different Retraining Methods vs Usual Care on the Prevention of Peritonitis in Peritoneal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Institute of Nephrology, Division of Renal, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PD TRAINING
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2019-07

CONDITIONS: Peritonitis
Keywords: peritoneal dialysis; retraining; peritonitis
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- operation inspection (Experimental): During retraining the patients performed bag exchange under the supervision of a nurse. The nurse ensured that each error listed in the NAC form should be avoided, thus immediately corrected any wrong steps if only.
  Interventions: Behavioral: operation inspection
- verbal education (Experimental): Patients in the oral education group also underwent retraining every 2 months. A nurse would address all items in the NAC form one by one, to remind the patient of the key points of bag exchange. Scores calculated by the sum of error items during the bag exchange for patients in technique inspection group, or by the sum of "yes" in the interactive quiz for patients in verbal education group.
  Interventions: Behavioral: operation inspection
- usual care (Experimental): Patients in the usual care group did not receive any retraining
  Interventions: Behavioral: operation inspection

INTERVENTIONS:
Behavioral: operation inspection — Retraining via operation inspection means that nurses check if patients can follow the taught skill during the procedure of bag exchange and correct wrong steps in one-to-one way every 2 months.
  Retraining via verbal education means that nurses remind patients of key points of bag exchange through interactive quiz derived from above checklist every 2 months till 24 months

SUMMARY:
To examine whether retraining via operation inspection or verbal education can reduce the risk for peritonitis in PD patients.

DETAILED DESCRIPTION:
The design is prospective, randomized, controlled study. At baseline (during the first month), they will receive a standard training program on performing bag exchange and education on the prevention of peritonitis.

Then the participants will be randomized into three groups: retraining via operation inspection (G1), retraining via verbal education (G2) and usual care (G3). Retraining will be performed every 2 months in G1 and G2 group.

During the following 2 years or a longer period, all the participants will be followed up frequently with outcome events recorded.

ELIGIBILITY:
Inclusion Criteria:

* CAPD patients.
* Medically stable and receiving PD for<1 week
* age between 18 and 80 years
* self-care or doing bag exchange by a fixed assistant Exclusion Criteria
* followed up at least every 2 months
* dialyzed with glucose lactate-buffered PD solutions produced by Baxter Corp, China

Exclusion Criteria:

* Pregnancy;
* undergoing APD therapy
* Intolerance to the study protocols;
* Severe and unstable condition, acute or chronic inflammation disease;
* a high probability (assessed by the recruiting physician) of receiving a kidney transplant or transferring to HD or drop-out due to socioeconomic causes within 6 months;
* suffering peritonitis before receiving the interventions
* cognitive or psychological dysfunction;
* communication barrier

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-12; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
first-episode peritonitis | 48 months
  Infection rates were calculated as the number of infections divided by the total time at risk, and expressed as episodes per 100 patient-years at risk.

SECONDARY OUTCOMES:
first-episode enteric peritonitis,first-episode non-enteric peritonitis | 48 moths
  Enteric organisms included enterococcus and enterobacter.
transition transition to haemodialysis, and all-cause death. | 48 moths
  transition to haemodialysis, and all-cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dong, MD,PhD,, Principal Investigator — Peking University First Hospital
Locations (1):
- Jie Dong, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu Y, Zhang Y, Yang B, Luo S, Yang Z, Johnson DW, Dong J. Prevention of peritoneal dialysis-related peritonitis by regular patient retraining via technique inspection or oral education: a randomized controlled trial. Nephrol Dial Transplant. 2020 Apr 1;35(4):676-686. doi: 10.1093/ndt/gfz238. PMID 31821491